CLINICAL TRIAL: NCT06218511
Title: A Phase I Trial of IMA970A Plus Montanide in Combination With Durvalumab (Anti-PD-L1) in Patients With Very Early, Early and Intermediate Stage of Hepatocellular Carcinoma After Any Standard Treatments
Brief Title: A Phase I Trial of IMA970A Plus Montanide in Combination With Durvalumab (Anti-PD-L1)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEPAVAC 201; 46/22 (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2023-10-30; First posted 2024-01-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; Monatide (IMS 3015); Adjuvants, Pharmaceutic

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): single-arm open-label
  Interventions: Biological: Peptide-based hepatocellular carcinoma vaccine IMA970A; Combination Product: Durvalumab; Other: Montanide (Adjuvant)

INTERVENTIONS:
Biological: Peptide-based hepatocellular carcinoma vaccine IMA970A — IMA970A is a lyophilized multi-peptide vaccine consisting of 17 individual peptides (active pharmaceutical ingredients) and 2 excipients (Poloxamer 338 and Mannitol). All peptides have been chemically manufactured by well established solid phase peptide synthesis procedures. All peptides are composed of linear, unmodified L- amino acid chains with chain length in the range of 9 to 21 amino acids.
Combination Product: Durvalumab — anti-PD-L1
Other: Montanide (Adjuvant) — Montanide ISA™ 51 is a water-in-oil (W/O) emulsion composed of a mineral oil and a surfactant from the mannide monooleate family with immune stimulatory effect .

SUMMARY:
The trial is designed as a single-arm, open-label, phase I study investigating an off-the-shelf, multi-peptide-base HCC vaccine plus Montanide, combined with Durvalumab in patients with very early, early and intermediate stage of HCC. The investigational agents will be applied without concomitant anti-tumour therapy with the intention to reduce risk of recurrence/progression in patients who have received all indicated standard treatments.

DETAILED DESCRIPTION:
The proposed phase I HepaVac-201 will investigate safety, tolerability and immunogenicity of the same investigational IMA-970A agent, formulated in Montanide combined with an anti-PD-L1 (i.e.Durvalumab). Compared to the previous HepaVac-101 clinical trial, two major differences are introduced. The adjuvant Montanide (oil and water mix) will replace the CV8102 (TLR agonist) which was used in the HepaVac-101 trial. The anti-PD-L1 Durvalumab is introduced in the protocol. Indeed, several reports have shown that, inhibitory receptors are induced after vaccination. Blocking these inhibitory pathways lead to amplification of the T cell-mediated immune response. In particular, IFNγ production by antitumour-specific T cells could also upregulate PD-L1 on tumour cells, as a resistance mechanism to adaptive immunity, thereby promoting PD-L1-PD-1 blockade after vaccination. Several early phases clinical trials have been performed to validate this hypothesis. The aim is to verify whether these two changes in the HepaVac-201 protocol will improve the immunogenicity of the vaccine keeping the same safety profile as in the HepaVac-101 protocol. The phase I clinical trial HepaVac-201 will be conducted at the Istituto Nazionale Tumori, IRCCS Fondazione G. Pascale, Naples, Italy. Dr. Luigi Buonaguro will be the coordinator of the trial. Dr. Francesco Izzo and Dr. Paolo A. Ascierto are the lead Investigators. The trial is designed as a single-arm, open-label, phase I study investigating an off-the-shelf, multi-peptide-base HCC vaccine plus Montanide, combined with Durvalumab in patients with very early, early and intermediate stage of HCC. The investigational agents will be applied without concomitant anti-tumour therapy with the intention to reduce risk of recurrence/progression in patients who have received all indicated standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age > 18 years at time of study entry.
3. HLA type: HLA-A*02 and/or HLA-A*24 positive.
4. Very early, early and intermediate stage (Barcelona Clinic Liver Cancer (BCLC) stage 0, A, B disease) hepatocellular carcinoma (HCC) diagnosed by biopsy or resected tissue (patho-histological diagnosis) or imaging findings (non-invasive criteria) following any standard treatment (e.g. hepatic resection, Radiofrequency Ablation / Percutaneous Ethanol injection (RFA/PEI), Transarterial chemoembolization (TACE) and SIRT) and without any evidence of active disease that warrant further treatment.
5. Minimum life expectancy of 1 year.
6. Patho-histological diagnosis of HCC based on biopsy is required for all nodules occurring in non-cirrhotic livers, and for those cases with inconclusive or atypical imaging appearance in cirrhotic livers.
7. Non-invasive criteria can only be applied to cirrhotic patients and need to be based on imaging techniques obtained by 4-phase multidetector CT scan or dynamic contrast enhanced MRI and on the identification of the typical hallmark of HCC (hypervascular in the arterial phase with washout in the portal venous or delayed phase). One imaging technique is sufficient for nodules beyond 1 cm (> 1 cm) in diameter.
8. Patients for whom no standard anti-tumour therapy is indicated for the next 3 months thereafter any standard anti-tumour therapies applied for the treatment of BCLC stage 0, A and B HCC (e.g. RFA/PEI, TACE, and SIRT) are allowed to be applied in combination with the study treatment. Patients for whom treatment for advanced disease (e.g.

   sorafenib) is indicated will be withdrawn from study treatment.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0/1 with the specific characteristics indicated in the exclusion criteria.
10. Child-Pugh A5-6 and B7 disease or no liver function impairment.
11. Body weight >30 kg.
12. Adequate normal organ and marrow function as defined below:

    1. Haemoglobin ≥9.0 g/dL
    2. Absolute neutrophil count (ANC) ≥1.0 × 109 /L
    3. Platelet count ≥75 × 109

       /L
    4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    5. AST (SGOT)/ALT (SGPT) ≤5 x institutional upper limit of normal
    6. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    Males:

    Creatinine CL (mL/min)

    = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min)

    = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
13. Willingness and ability to comply with the study protocol for the duration of the study.
14. Female patient of child-bearing potential:

    * Female patients of childbearing potential who are not totally sexually abstinent (i.e., refraining from heterosexual intercourse during the entire period of risk associated with study interventions) and intend to be sexually active with a non sterilised male partner must use at least 1 highly effective method of contraception (Appendix 4). They should have been stable on their chosen method of birth control for a minimum of 3 months before entering the study and continue to use it throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of study treatment). Non sterilised male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period.

Male patients with a female partner of childbearing potential:

* Non-sterilised male patients who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of study treatment). Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period. Vasectomised males are considered fertile and should still use a male condom plus spermicide as indicated above during the clinical study.
* Even if the female partner is pregnant, male participants should still use a condom plus spermicide (where approved), as indicated above during the clinical study, if there is a concern about damaging the developing foetus from drug in ejaculate.
* Female partners (of childbearing potential) of male patients must also use a highly effective method of contraception throughout this period (Appendix 4).

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Any prior systemic anti-tumour treatment (including drug or treatment regimen, approved or experimental) within 2 weeks before study treatment administration.
2. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable
3. Liver transplanted patients; patients who are on the liver transplantation waiting list are not allowed to be enrolled.
4. Concurrent enrolment in another clinical study, unless it is an observational (non interventional) clinical study or during the follow-up period of an interventional study.
5. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
6. History of allogenic organ transplantation.
7. History or evidence of systemic autoimmune disease, e.g. rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus (SLE), scleroderma, Sjögren's syndrome, Wegener's granulomatosis, Guillain-Barre syndrome.
8. Need for concomitant treatment with immunosuppressive drugs or other immune modifying drugs. The use of inhaled and nasally applied steroids, as well as topical steroids outside the vaccination area are permitted.
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
10. History of other malignancies within the last 3 years except for adequately treated except cervical carcinoma in situ, basal cell carcinoma and superficial bladder tumours [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to signing of informed consent by the patient.
11. History of leptomeningeal carcinomatosis.
12. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart). Regardless of whether this criterion stays or not, all patients should have a baseline ECG.
13. Any medically diagnosed or suspected condition of immunodeficiency or medical history thereof
14. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
15. Any other known infection with a biological agent that can cause a severe disease and poses a severe danger to lab personnel working on patients' blood or tissue.

    Examples are: rabies, Mycobacterium leprae, Plasmodium falciparum, Coccidioides immitis.
16. Acute and active infections requiring oral or intravenous antibiotics, antiviral or antifungal therapy within 30 days prior to enrolment (exception: Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infections; direct-acting antivirals may be applied as medically indicated).
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note:

    Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 6 months after receiving the last dose of treatment combination or 3 months after receiving the last dose of durvalumab monotherapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
21. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

    1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to be enrolled if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    4. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

       * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection
       * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
       * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
22. Patients undergoing renal dialysis or with relevant chronic renal failure.
23. Abnormal laboratory values as specified below:

    1. Haematology: Haemoglobin (< 8.5 g/dL), platelets (< 75,000/μL), leukocytes (< 2,500/μL), neutrophils (< 1,000/μL), lymphocytes (< 500/μL)
    2. Liver function: serum bilirubin (≥ 3 x ULN), Alanine aminotransferase (ALAT) or Aspartate aminotransferase (ASAT) (≥ 5 x ULN)
    3. Renal function: serum creatinine (≥ 1.5 x ULN)
24. Patients with seizure disorder requiring medication (such as steroids or anti epileptics drugs).
25. Encephalopathy.
26. Clinically relevant ascites with the only exception of patients that remain free from symptomatic ascites under low-dose diuretics (Spironolactone >100 mg daily and Furosemide >40 mg daily).
27. Hypersensitivity to the study drugs (IMA970A, Montanide or Durvalumab) including excipients and to CT/MRI contrast agent.
28. Evidence of current alcohol or drug abuse.
29. Serious intercurrent illness, which according to the investigator, poses an undue risk to the patient when participating in the trial, including, but not limited to, any of the following:

    1. Clinically significant cardiovascular disease (e.g., uncontrolled hypertension; clinically significant cardiac arrhythmia, clinically significant QT-prolongation)
    2. New York Heart Association class III-IV congestive heart failure
    3. Symptomatic peripheral vascular disease
    4. Severe pulmonary dysfunction
    5. Psychiatric illness or known social situation that would preclude study compliance
    6. Systemic inflammatory condition
30. Less than 6 months since any of the following:

    1. Myocardial infarction
    2. Severe or unstable angina pectoris
    3. Coronary or peripheral artery bypass graft
    4. Cerebrovascular event incl. transient ischemic attack
    5. Pulmonary embolism / deep vein thrombosis (DVT)
31. Any condition which in the judgment of the investigator would place the patient at undue risk or interfere with the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 55 months (approximately 4.5 years)
  Safety assessments will consist of continuous monitoring and reporting of adverse events (AEs) including serious adverse events (SAEs), regular monitoring of vital signs, ECOG performance status and regular conduct of physical examinations and laboratory assessments (haematology, clinical [bio]chemistry including C reactive protein (CRP) and glomerular filtration rate (GFR), coagulation test, assessment of viral infection, thyroid function test (TFT), urinalysis), electrocardiogram (ECG) and pregnancy tests (if applicable). Possible cross-reactivity with live attenuated vaccination or flu vaccine will be assessed.

SECONDARY OUTCOMES:
Additional immunological parameters in blood (e.g. regulatory T-cells, myeloid derived suppressor cells) | 55 months (approximately 4.5 years)
  The number of events and the frequency of several MDSC and Treg populations will be presented.
Infiltrating T-lymphocytes, immune cells and potential other (bio)markers in tumour tissue (depending on availability of tissue) | 55 months (approximately 4.5 years)
  The number of events and the frequency of infiltrating T-lymphocytes (TILs), other immune cells and potential other (bio)markers will be presented.
DFS | 55 months (approximately 4.5 years)
  Disease-free survival
PFS | 55 months (approximately 4.5 years)
  progression-free survival
OS | Patients will be followed for overall survival every 2 months for up to 2 years after having completed the interventional part of the study at EOS.
  Overall survival

OTHER OUTCOMES:
Immunogenicity | 55 months (approximately 4.5 years)
  The assessment of T-cell response in peripheral blood will be performed for all patients using standardized immune-monitoring assays. Peripheral blood mononuclear cells (PBMCs) of patients will be analysed for the occurrence of T-cell responses to peptides contained in IMA970A vaccine before application of standard therapy, such as before and after vaccination. The induction of immune responses by IMA970A vaccine will be subsequently analysed.
Additional immunological parameters | 55 months (approximately 4.5 years)
  e.g. regulatory T-cells, myeloid-derived suppressor cells
Infiltrating T-lymphocytes in tissue | 55 months (approximately 4.5 years)
  Infiltrating T-lymphocytes in tissue (depending on availability of tissue)
Serum/plasma biomarkers | 55 months (approximately 4.5 years)
  Analysis of other immune cell populations that may influence T-cell responses such as regulatory T cells (Tregs) and myeloid-derived suppressor cells (MDSC) (cellular biomarkers) will be performed using PBMCs from pre- and post-vaccination time points.
Assessment of the potential impact of the standard therapy on the natural immune response to peptides contained in IMA970A | 55 months (approximately 4.5 years)
  The assessment of the natural immune response to peptides contained in IMA970A will be performed before start of standard anti-tumor therapy and thereafter (S 2) to assess whether the selected standard therapy has an influence on a potentially pre-existing (natural) immune response. Thus, available blood samples are used to reach this study endpoint and can therefore be justified, even if some patients turn out not to be eligible for study participation during S 2 procedures. Standardized sample collection, PBMC isolation and storage and standardized immunomonitoring assays will be used for this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Antonio Ascierto, Principal Investigator — IRCCS I.N.T. "G. Pascale"; Francesco Izzo, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (1):
- Luigi Buonaguro, Napoli, Napoli, Italy